CLINICAL TRIAL: NCT04672525
Title: Rifabutin Versus Rifampicin for Treatment of Staphylococcal Prosthetic Joint Infection Treated With Debridement, Antibiotics and Implant Retention (DAIR Strategy): a Multicenter Randomized, Open-label, Non-inferiority Trial
Brief Title: Rifabutin Versus Rifampicin for Treatment of Staphylococcal PJI Treated With DAIR
Acronym: RIFAMAB
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIPH_2019_01
Record Dates: First submitted 2020-10-11; First posted 2020-12-17 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Prosthetic Infection
MeSH Terms: interventions — Rifabutin; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIFAMPICIN (Active Comparator): Patient with staphylococcal PJI, treated with DAIR strategy, and randomized in the control group will receive rifampicin in association with another antibiotic except rifabutin, as-per recommendations for 12 weeks.
  Interventions: Drug: Rifampicin
- RIFABUTIN (Experimental): Patient with staphylococcal PJI treated with DAIR strategy, and randomized in the experimental group, will receive rifabutin in association with another antibiotic except rifampicin, as-per recommendations for 12 weeks.
  Interventions: Drug: Rifabutin

INTERVENTIONS:
Drug: Rifabutin — 2 tablets of 150 mg per day rifabutin tablet daily for 12 weeks in 1 administration with a companion treatment
  Arms: RIFABUTIN
Drug: Rifampicin — 10 mg/kg per day (range 600 mg to 1,200 mg) rifampicin tablet in 1 daily dose for 12 weeks with a companion treatment
  Arms: RIFAMPICIN

SUMMARY:
Rifampicin, is key in the treatment of staphylococcal PJIs. Rifabutin has a better profile of tolerance than rifampicin regarding the risk of interaction with concomitant medications and liver disorders. The hypothesis is that rifabutin may be an alternative antibiotic option as efficient as rifampicin for the treatment of staphylococcal PJIs, with a better safety profile. The investigator aim to demonstrate the non-inferiority of rifabutin as compared with rifampicin prescribed in combination treatment for PJIs.

ELIGIBILITY:
Inclusion Criteria:

1. Hip or knee Prosthetic joint infection treated by debridement, antibiotic therapy initiation and retention of prothesis (DAIR strategy)
2. Infected with at least one of the following microorganisms:

   1. Staphylococcus aureus
   2. Coagulase-negative staphylococci
3. Microorganisms susceptible to rifampicin and at least one other antibiotic suitable for the treatment of PJI (e.g., penicillin, fluoroquinolone, (doxy/mino)cycline, oxazolidinone, cotrimoxazole, daptomycin, glycopeptide, macrolide, fusidic acid), regardless of sensitivity to methicillin.
4. Age ≥ 18 years
5. At least 2 days of appropriate (i.e., covering pathogen(s) identified in the intraoperative samples) empirical agents are needed. Pre-randomization antimicrobial therapy could be: flucloxacillin, oxacillin, vancomycin, daptomycin. β-lactam plus β-lactamase-inhibitors (e.g. ampicillin+sulbactam, piperacillin+tazobactam), cephalosporins (except ceftazidime), carbapenems, teicoplanin, ceftaroline, ceftobiprole.
6. Signed Inform consent
7. Patient having the rights to French social insurance
8. For women of childbearing potential i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile and excluding oestroprogestative-based contraception, any effective contraceptive: vasectomy (for men), intrauterine device copper, feminine sterilization, condom, sexual abstinence is required. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause

Exclusion Criteria:

1. Suspicion of reduce absorption of oral treatment due to abdominal disorder Known or suspected malabsorption (imperfect absorption of food material by the small intestine)
2. Polymicrobial infection due to other than staphylococcus species susceptible to rifampicin
3. Known or suspected allergy to rifabutin and/or rifampicin
4. Diagnosis of endocarditis associated to PJI
5. Renal transplant or Chronic kidney disease with an eGFR of less than 30ml/min/1.73m²
6. Other Solid Organ Transplant
7. Liver cirrhosis, Child-Pugh score C
8. Any other concomitant infection which required a prolonged course of intravenous antibiotic therapy
9. Oestroprogestative-based contraception
10. Oral anticoagulant drugs
11. Other drug-drug interaction that contraindicated rifampicin or rifabutin
12. Porphyria
13. Unable to take oral treatment
14. Receive empirical postoperative antibiotic treatment by rifampicin or rifabutin prior to randomization
15. Pregnancy or lactating women
16. Curator or guardianship or patient placed under judicial protection
17. Participation in other interventional research during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | At one year
  Treatment failure defined as one of following events:
  * The need for any further surgical procedure - i.e. implants removal, implants exchange or amputation;
  * And/or PJI related death;
  * And/or use of suppressive antibiotic therapy that was not planned before randomization

SECONDARY OUTCOMES:
Occurrence of serious adverse events (SAEs), including death (i.e. all cause) | At the end of 12 weeks duration of antibiotic treatment planned
  Proportion of patient which are free from SAEs occurrence, as defined by:
  -Patients who completed the entire 12 weeks duration of antibiotic treatment planned initially and; xWho did not experience grade 3-4 adverse events, including death, regardless of the link with antibiotic therapy; xWho did not experience adverse events which led to either to:
  * Reduce the dosage or split the treatment to two take/day;
  * Or stop any component of the antibiotic treatment.
Occurrence of any adverse event that could be related to rifampicin or rifabutin | At the end of 12 weeks duration of antibiotic treatment planned
  Number and rate of patients in each arm who experiences:
  * Liver cytolysis (>=2N for ALT AND/OR AST)
  * Acute Kidney failure as defined by serum creatinine increase in KDIGO
  * Digestive symptoms, including diarrhea
  * Who required a modification of antibiotic dosage during the 12 weeks' period of antibiotic treatment
  * Uveitis/ophthalmologic disorder
  * Neurological disorder
Proportion of patients from each arm who will complete the 12-week duration of rifampicin/rifabutin treatment, early termination of the planned 12 weeks' period of antibiotics | At the end of 12 weeks duration of antibiotic treatment planned
  Early termination rate will be measured in each arm, as the number of patients having stopped rifampicin or rifabutin before the planned 12 weeks period over the total number of patients enrolled in the studied arm.
Adherence to antibiotics regimen | At the end of 12 weeks duration of antibiotic treatment planned
  Adherence rate to medication will be measured as the number of days on which all doses were missed over the number of days of planned antibiotic therapy. Patients enrolled in the study will have to fill their pill count in a daily notebook.
Quality of life, as evaluated by EQ 5D 3L questionnaire | At the end of the study follow up, an average of 24 months
  Quality of life, as evaluated by the use EQ 5D 3L auto-questionnaire as used in previous randomized clinical trial on bone and joint infection
Functional prognosis using Oxford questionnaire evolution according to location of PJI | At the end of the study follow up, an average of 24 months
  Oxford Scores as used in previous randomized clinical trial on bone and joint infection
Long term efficacy of rifampicin and rifabutin treatment | At the end of the study follow up, an average of 24 months
  Long term efficacy: treatment failure, as defined for primary outcome, at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric SENNEVILLE, Md PhD, Principal Investigator — CH TOURCOING
Locations (30):
- France (30):
  - CHU Amiens Picardie, Amiens
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - CH de Béthune, Béthune
  - CHU Bordeaux, Bordeaux
  - APHP Hôpital Ambroise Paré, Boulogne-Billancourt
  - CHRU Brest, Brest
  - CHU Caen, Caen
  - CH Alpes Leman, Contamine-sur-Arve
  - CHU Dijon Bourgogne, Dijon
  - CHU Grenoble Alpes, Grenoble
  - CHRU Lille, Lille
  - GHICL Hôpital Saint Vincent de Paul, Lille
  - CHU de Limoges, Limoges
  - GHICL Hôpital Saint Philibert, Lomme
  - Clinique de la Sauvegarde, Lyon
  - Hospices Civils de Lyon, Lyon
  - APHM Hôpital Nord, Marseille
  - CHU Nice, Nice
  - CH Annecy Genevois, Pringy
  - CH Cornouaille, Quimper
  - CHU Reims, Reims
  - CHU de Rennes, Rennes
  - CHU Saint Etienne, Saint-Priest-en-Jarez
  - CHRU Strasbourg, Strasbourg
  - Hôpital d'instruction des armées Sainte Anne, Toulon
  - Clinique Joseph Ducuing, Toulouse
  - Clinique Médipole Garonne, Toulouse
  - CH Tourcoing, Tourcoing
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: No